CLINICAL TRIAL: NCT01063686
Title: Use of a Cervical Cap as an Aid in Uncertain Rupture of Membranes in the Second Trimester
Brief Title: The Cervical Cap in the Diagnosis of Rupture of Membranes in the Second Trimester
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Funding
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, david danon, Doctor, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: rmc-0191
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Fetal Membranes, Premature Rupture; Ultrasonography
Keywords: Pregnancy
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Insemination cervical cap (No Intervention)
  Interventions: Device: insemination cervical cap

INTERVENTIONS:
Device: insemination cervical cap — Primary abdominal ultrasound (US) for amniotic fluid index (AFI), Single vertical pocket, and dimensions of pocket below the presenting part. Speculum vaginal examination. In a sterile manner a cervical cap is adjusted on the cervix. the patient is kept recumbent for 6 hours. A repeat US exam is performed. The cervical cap is removed. After one hour another US is performed.
  Other Names: CERVICAL CUP pre-cut standard size, C.C.D. International.; Ref. 12050IS; 48, rue des Petites Ecuries; 75010 Paris; France

SUMMARY:
Early preterm premature rupture of membranes (PPROM) complicates 0.7% of pregnancies. When PPROM occurs before the 24th week,the risk of fetal and neonatal death is 70%. There is also a high risk of neonatal and maternal morbidity. When the diagnosis of PPROM is uncertain by physical examination, additional tests are needed. These tests have false positive and false negative rates. The gold standard for diagnosing PPROM is amniocentesis and dye test. This procedure has a risk of infection and abortion.Our hypothesis is that by using a cervical cap for 6 hours and repeated ultrasound exams we can diagnose or rule out PPROM in cases which are uncertain. Our study group will be pregnant women gestational age 14-23, suspected of having PPROM.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 14-23
* Single fetus
* Suspected rupture of membranes
* Oligohydramnios

Exclusion Criteria:

* Vaginal bleeding
* Suspected chorioamnionitis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Changes in amniotic fluid index and single vertical pocket before and after placement of the cervical cap/ | the parameters will be measured before placement, 6 hours after placement, 1 hour after displacement

SECONDARY OUTCOMES:
chorioamnionitis and abortion | one week from the start of the study

CONTACTS AND LOCATIONS:
Overall Officials: David Danon, MD, Principal Investigator — Department of Ob/Gyn Rabin Medical Center, Israel
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel